CLINICAL TRIAL: NCT01571609
Title: Baseline Physiology Studies in Carriers of Gene Variant X Conferring Major Risk of CVD-prone Metabolic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Lundbeck Foundation (Other); Aarhus University Hospital (Other); Vejle Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Steno Diabetes Center Copenhagen (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Julie Støy, MD, University of Aarhus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1-10-72-113-12
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Hyperlipidemia; Diabetes Mellitus; Metabolic Syndrome; Arterial Hypertension; Obesity
MeSH Terms: conditions — Hyperlipidemias; Diabetes Mellitus; Metabolic Syndrome; Hypertension; Obesity | interventions — NDC80 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carriers (Experimental)
  Interventions: Other: first phase insulin secretion (FPIR), Hyperinsulinemic euglycemic clamp (HEC), glucose tracer, and palmitate tracer
- Non-carriers (Experimental)
  Interventions: Other: first phase insulin secretion (FPIR), Hyperinsulinemic euglycemic clamp (HEC), glucose tracer, and palmitate tracer

INTERVENTIONS:
Other: first phase insulin secretion (FPIR), Hyperinsulinemic euglycemic clamp (HEC), glucose tracer, and palmitate tracer — FPIR: intravenous infusion of 20 % glucose 0.3 mg/kg in 2 minutes followed by blood sampling at times 0, 2, 4, 6, 8, and 10. Duration 10 minutes.
  HEC: intravenous infusion of actrapid 1mU/kg/minute, simultaneous infusion of 20 % glucose at variable rate to reach plasma blood glucose level of 5 mmol/L. Duration 120 minutes
  Glucose tracer: bolus of 3H3glucose (12µCi) followed by infusion of 3H3glucose (0,12 µCi/min). Duration 120 minutes.
  Palmitate tracer:[9,10-3H]-palmitate 0,3 µCi/min. Duration 60 minutes.

SUMMARY:
The purpose of the present study is to conduct a thorough and relevant physiology study of carriers and non-carriers of the gene variant X in order to determine the effect of the genetic variant on various metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-70 years of age
* Member of Biobank Vejle
* BMI<30

Exclusion Criteria:

* Diabetes mellitus
* Severe illness

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
insulin secretion | 10 minutes
  Estimation of first phase insulin secretion

SECONDARY OUTCOMES:
Insulin resistance | 240 minutes
  Estimation of insulin resistance using hyperinsulinemic euglycemic clamp and glucose and lipid tracers
body composition | 60 minutes
  Evaluation of body composition using Dxa scan and MRI scan
atherosclerosis | 30 minutes
  Evaluation of presence and severity of atherosclerosis using ultrasound scan of the common carotide artery
biochemical blood profiling | at baseline
  Various tests run on blood samples
Insulin resistance | 60 minutes
  Biopsi from muscle and adipose tissue performed at baseline and during clamp study.
Blood pressure | 24 hours
  Measurement of blood pressure every 20. minutes/24 hours
Indirect calorimetry | 60 minutes
  Estimation of resting energy expenditure and respiratory quotient

CONTACTS AND LOCATIONS:
Overall Officials: Niels Møller, Professor, Principal Investigator — University of Aarhus; Oluf B Pedersen, Professor, Principal Investigator — Steno Diabetes Center Copenhagen; Torben Hansen, Professor, Principal Investigator — Steno Diabetes Center Copenhagen; Jørgen Rungby, Professor, Principal Investigator — University of Aarhus
Locations (1):
- Medicinsk forskningslaboratorium, Aarhus Universitet, Aarhus, Denmark

REFERENCES:
- [Derived] Stoy J, Kampmann U, Mengel A, Magnusson NE, Jessen N, Grarup N, Rungby J, Stodkilde-Jorgensen H, Brandslund I, Christensen C, Hansen T, Pedersen O, Moller N. Reduced CD300LG mRNA tissue expression, increased intramyocellular lipid content and impaired glucose metabolism in healthy male carriers of Arg82Cys in CD300LG: a novel genometabolic cross-link between CD300LG and common metabolic phenotypes. BMJ Open Diabetes Res Care. 2015 Aug 26;3(1):e000095. doi: 10.1136/bmjdrc-2015-000095. eCollection 2015. PMID 26336608
- [Derived] Stoy J, Grarup N, Horlyck A, Ibsen L, Rungby J, Poulsen PL, Brandslund I, Christensen C, Hansen T, Pedersen O, Moller N, Kampmann U. Blood pressure levels in male carriers of Arg82Cys in CD300LG. PLoS One. 2014 Oct 14;9(10):e109646. doi: 10.1371/journal.pone.0109646. eCollection 2014. PMID 25314291
- See also: Project home page — http://lucamp.org